CLINICAL TRIAL: NCT04817995
Title: Stress Recovery Program FOREST for Healthcare Staff: A Randomized Controlled Trial
Brief Title: Stress Recovery Program FOREST for Healthcare Staff
Acronym: FOREST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Evaldas Kazlauskas, Professor, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-03-22/61
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Perceived Stress
Keywords: Healthcare staff; Perceived stress; Internet intervention; Recovery; Efficacy
MeSH Terms: interventions — Forests

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated either to the intervention or control groups. The control group is a waiting list. The control group will participate in the intervention after it will be completed for the intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will get a 6-week internet-based stress recovery intervention.
  Interventions: Behavioral: FOREST
- Control group (No Intervention): The waiting list will get no intervention while the intervention group is getting the intervention. The waiting list has the possibility to get an intervention after the intervention group finishes it.

INTERVENTIONS:
Behavioral: FOREST — Intervention is going to take the form of an internet-based stress recovery intervention consisting of six modules. The themes include introduction, psychological detachment, distancing, mastery, control, and keeping the change alive. These themes were chosen after considering topics that might be the most useful for healthcare staff experiencing high levels of stress. Each module consists of psychoeducation and exercise parts. Psychologist provide individual feedback on completed exercises as well as can be reached on demand.
  Arms: Intervention group

SUMMARY:
The aim of the study is to assess the efficacy of an internet-based stress recovery intervention among healthcare staff during COVID-19 pandemic.

DETAILED DESCRIPTION:
Intervention is going to take the form of an internet-based stress recovery intervention consisting of six modules. The themes include introduction, psychological detachment, distancing, mastery, control, and keeping the change alive. These themes were chosen after considering topics that might be the most useful for healthcare staff experiencing high levels of stress. Each module consists of psychoeducation and exercise parts. Psychologist provide individual feedback on completed exercises as well as can be reached on demand.

The effect of the intervention will be compared against a waiting list control group. Intervention is in Lithuanian.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old;
* comprehending Lithuanian language;
* access to internet;
* high levels of stress.

Exclusion Criteria:

* acute psychiatric crisis;
* high suicide risk;
* interpersonal violence;
* alcohol / drug addiction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change on Recovery Experience Questionnaire | Pre-treatment, after 6 weeks, 3 months post-treatment
  Changes on stress recovery are measured. Recovery Experiences Questionnaire (Sonnentag & Fritz, 2007) is a self-report measure and consists of 16 questions. All items are answered on a 5-point Likert scale that ranges from 1 (Totally disagree) to 5 (Totally agree). Higher score indicates more pronounced recovery.

SECONDARY OUTCOMES:
Change on International Trauma Questionnaire | Pre-treatment, after 6 weeks, 3 months post-treatment
  Changes on post-traumatic stress disorder are measured. International Trauma Questionanaire (ITQ, Cloitre et al., 2018) is a self-report measure and consists of 18 questions. All items are answered on a 5-point Likert scale that ranges from 0 (not at all) to 4 (extremely). Higher score indicates more pronounced symptoms.
Change on Moral Injury Outcome Scale | Pre-treatment, after 6 weeks, 3 months post-treatment
  Changes on moral injury are measured. Moral Injury Outcome Scale (MIOS, Litz et al., 2020) is a self-report measure and consists of 15 questions. All items are answered on a 5-point Likert scale that ranges from 0 (Strongly disagree) to 4 (Strongly agree). Higher score indicates more pronounced moral injury.
Change on Perceived Stress Scale | Pre-treatment, after 6 weeks, 3 months post-treatment
  Changes on perceived stress are measured. Perceived Stress Scale (PSS-4, Cohen et al., 1983) is a self-report measure and consists of 4 questions. All items are answered on a 5-point Likert scale that ranges from 0 (Never) to 4 (Very often). Higher score indicates more pronounced perceived stress.
Change on Patient Health Questionnaire | Pre-treatment, after 6 weeks, 3 months post-treatment
  Changes on depression and anxiety are measured. Patient Health Questionnaire-4 (PHQ-4, Kroenke et al., 2009) is a self-report measure and consists of 4 questions. All items are answered on a 4-point Likert scale that ranges from 0 (Not at all) to 3 (Nearly every day). Higher score indicates more pronounced depression and anxiety.
Change on Well-being Index | Pre-treatment, after 6 weeks, 3 months post-treatment
  Changes on well-being are measured. Well-being Index (WHO-5, Bech, 2004) is a self-report measure and consists of 5 questions. All items are answered on a 6-point Likert scale that ranges from 0 (At no time) to 5 (All of the time). Higher score indicates more pronounced well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Vilnius University, Vilnius, Lithuania

REFERENCES:
- [Derived] Dumarkaite A, Truskauskaite I, Andersson G, Jovarauskaite L, Jovaisiene I, Nomeikaite A, Kazlauskas E. The efficacy of the internet-based stress recovery intervention FOREST for nurses amid the COVID-19 pandemic: A randomized controlled trial. Int J Nurs Stud. 2023 Feb;138:104408. doi: 10.1016/j.ijnurstu.2022.104408. Epub 2022 Nov 24. PMID 36527859
- [Derived] Jovarauskaite L, Murphy D, Truskauskaite-Kuneviciene I, Dumarkaite A, Andersson G, Kazlauskas E. Associations between moral injury and ICD-11 post-traumatic stress disorder (PTSD) and complex PTSD among help-seeking nurses: a cross-sectional study. BMJ Open. 2022 May 9;12(5):e056289. doi: 10.1136/bmjopen-2021-056289. PMID 35534083
- [Derived] Jovarauskaite L, Dumarkaite A, Truskauskaite-Kuneviciene I, Jovaisiene I, Andersson G, Kazlauskas E. Internet-based stress recovery intervention FOREST for healthcare staff amid COVID-19 pandemic: study protocol for a randomized controlled trial. Trials. 2021 Aug 21;22(1):559. doi: 10.1186/s13063-021-05512-1. PMID 34419114